CLINICAL TRIAL: NCT05364723
Title: Place of Glycation in Diabetic Retinopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mohammed VI University Hospital (Other)
Responsible Party: Principal Investigator, Oujidi Wissale, ophthalmology resident, Mohammed VI University Hospital
Other Study IDs: MohammedVIUHophtalmology
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Descriptor
Keywords: glycation; diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:  — no intervention

SUMMARY:
1. Definition: Diabetic retinopathy is a microangiopathic complication of diabetes diabetes mellitus. Its pathophysiology includes glycation and intracellular hypoxia. Diabetic retinopathy (DR) is a microvascular complication of diabetes. It is the leading cause of It is the leading cause of blindness and visual impairment in people under the age of 60 in industrialized countries.

   Chronic hyperglycemia during diabetes plays a major role in the occurrence of diabetic diabetic retinopathy by promoting protein glycation and the accumulation of glycation end products (GTPs). GTPs are a heterogeneous group of compounds resulting from non-enzymatic and irreversible reactions between reducing sugars and amine groups of biological molecules such as proteins, lipids or nucleic acids.
2. Interest: The aim of our work is to describe the mechanisms by which glycation participates in the pathophysiology of diabetic retinopathy and to discuss the use of AGEs as biomarkers in this biomarkers in this pathological context and the therapeutic means that limit the toxicity of of AGEs.

The study is designed through a retrospective and prospective observational study to establish the of glycation in the occurrence of diabetic retinopathy. It will describe the demographic demographic profiles, glycemic control, clinical and paraclinical status of patients with diabetic diabetic retinopathy and will evaluate the relationship between glycation and diabetic retinopathy as well as the factors that influence this glycation in these patients, and induce the occurrence and / or of diabetic retinopathy. The data collected will allow to improve the knowledge, the diagnosis and the treatment of diabetic diabetic retinopathy, as well as a good management of the patients who should benefit from a more individualized and individualized and adequate treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients type 1 and type 2, of both sexes, and of all ages. Regular follow-up

Exclusion Criteria:

* Other types of diabetes. Irregular follow-up.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: diabetic population in the eastern region of Morocco
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
distribution of diabetic retinopathy in eastern morocco | 1year

IPD SHARING:
Plan to Share IPD: No